CLINICAL TRIAL: NCT03153020
Title: Determinants of Adherence to Post-stroke/Transient Ischemic Attack Secondary Prevention Treatment: Cohort Study in the Rhône
Acronym: OBSTACLE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0037
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of patients with stroke or transient ischemic attack: The cohort will be constituted of all consecutive patients admitted for a stroke or transient ischemic attack by the Rhône's emergency medical help service (SAMU), or in one of the emergency unit or stroke unit of the Rhône area, and presenting a symptom-onset (the last time the patient was seen without deficit) less than 24 hours.
  Interventions: Other: Patients with stroke or transient ischemic attack

INTERVENTIONS:
Other: Patients with stroke or transient ischemic attack — Determination of factors associated to the conformity to secondary prevention treatment 1, 2 and 3 years post a stroke or transient ischemic attack.

SUMMARY:
The effectiveness of emergency management of acute ischemic stroke has improved considerably in recent years with thrombolysis and more recently thrombectomy. This improvement is accompanied by an increase in the number of stroke survivors. One of the major issues for these ever-increasing survivors is the prevention of recurrence. According to data from the 3 French registries, more than 20% of patients have at least one recurrence. Secondary prevention treatment has demonstrated his efficacy to prevent stroke recurrence.

This evolution justifies identifying factors associated with adherence to secondary prevention treatment, measured at 1 year post-stroke / transient ischemic attack (TIA), in patients included in the STROKE 69 cohort.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients treated for a stroke suspicion at the acute phase,
* with symptom onset (the last time the patient was seen without deficit ) less than 24 hours,
* Managed by the Rhône's emergency medical help service (SAMU), in one of the emergency unit or stroke unit of the Rhône area
* Having given their written consent for the extraction of their healthcare consumption data from the Health Insurance databases

Exclusion Criteria:

* Hemorrhagic stroke,
* Patient institutionalized in the year following the stroke / transient ischemic attack,
* Patient unable to take treatment alone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke or transient ischemic attack of the Rhone area
Sampling Method: Non-Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Compliance to secondary prevention treatment 1 year post a stroke or transient ischemic attack | 1 year post a stroke or transient ischemic attack
  The overall medication possession ratio is the average of the medication possession ratio calculated for each therapeutic class (antiplatelet agents, anticoagulants, antihypertensives, hypolipidemic agents and oral antidiabetics).
  The medication possession ratio will be calculated from dispensing data from regional health insurance database and prescription data from the STROKE 69 study. For each patient, a medication possession ratio (CMA7 index) will be obtained by the ratio of the quantity of medication units dispensed to the quantity of medication units prescribed.
Determination of factors influencing compliance with secondary prevention treatment 1 year post a stroke or transient ischemic attack | 1 year post a stroke or transient ischemic attack
  A phone call will be made to patients 1 year post a stroke or transient ischemic attack.
  The following determinants will be studied in the 5 dimensions defined by World Health Organization:
  1. Socio-economic: level of education, profession, health insurance
  2. Patient and family-social environment: age, sex, marital status, lifestyle, level of patient support in the management of their treatment, representation of the disease and beliefs about medication
  3. Care pathway: management of stroke / TIA in emergency or neurovascular unit, admission to rehabilitation unit, medical consumption and therapeutics acts in the year following stroke / TIA
  4. Pathology: TIA or ischemic stroke, duration of hospitalization in acute phase and type of hospital, history of stroke or TIA, disability and autonomy, fatigue, anxiety and depression, comorbidities
  5. Treatments: therapeutic class and number of treatments / polymedication.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Pôle Information Médicale Evaluation Recherche, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoarau D, Ramos I, Termoz A, Fernandez V, Rambure M, Allemann SS, Derex L, Haesebaert J, Schott AM, Viprey M. Determinants of adherence to post-stroke/transient ischemic attack secondary prevention medications: A cohort study. Eur J Neurol. 2024 Oct;31(10):e16395. doi: 10.1111/ene.16395. Epub 2024 Jul 2. PMID 38953278